CLINICAL TRIAL: NCT06568952
Title: Right Ventricular Function of Patients With Multiple Myeloma Treated With Carfilzomib
Brief Title: Right Ventricular Function in Patients Taking Carfilzomib
Status: Completed | Type: Observational
Sponsor: Central Hospital, Nancy, France (Other)
Responsible Party: Sponsor
Other Study IDs: 2023PI0512
Record Dates: First submitted 2024-08-20; First posted 2024-08-23 (Actual); Last update posted 2024-08-23 (Actual); Status verified 2023-12

CONDITIONS: Pulmonary Hypertension
MeSH Terms: conditions — Hypertension, Pulmonary

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Patients treated for multiple myeloma in the second line with carfilzomib may develop pulmonary hypertension. This is well documented in the literature. However, there are no studies looking at right ventricular function in these patients, both before and during treatment.

DETAILED DESCRIPTION:
Patients treated for multiple myeloma in the second line with carfilzomib may develop pulmonary hypertension. This is well documented in the literature. However, there are no studies looking at right ventricular function in these patients, both before and during treatment.

Patients had a cardiac ultrasound scan prior to the introduction of carfilzomib and an ultrasound scan following the introduction of carfilzomib. We will look at the evolution of right ventricular function parameters in these patients.

ELIGIBILITY:
Inclusion Criteria:

* Patients treated for multiple myeloma with carfilzomib
* Patients with echocardiogram before and under treatment.

Exclusion Criteria:

* /

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients with multiple myeloma treated with carfilzomib
Sampling Method: Probability Sample
Enrollment: 36 (Actual)
Dates: Start 2024-04-30 (Actual); Primary Completion 2024-06-30 (Actual); Study Completion 2024-07-30 (Actual)

PRIMARY OUTCOMES:
tricuspid annular plane systolic excursion | 6 months after carfilzomib treatment
  measurement of tricuspid annular plane systolic excursion by echocardiography

CONTACTS AND LOCATIONS:
Overall Officials: Simon Valentin, MD, Principal Investigator — Université de Lorraine, Département de Pneumologie, CHRU NANCY
Locations (1):
- Simon VALENTIN, Nancy, France

IPD SHARING:
Plan to Share IPD: No